CLINICAL TRIAL: NCT06398769
Title: Comparison of VCare and SecuFix Uterine Manipulator in Total Laparoscopic Hysterectomy
Brief Title: VCare Versus SecuFix Uterine Manipulator for Total Laparoscopic Hysterectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Esra Keles, Assoc Prof, MD, PhD candidate, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Device Feasibility
Other Study IDs: uterinemanipulator-1
Record Dates: First submitted 2024-04-26; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Operative Time; Length of Hospital Stay; Perioperative Complications
Keywords: uterine manipulator; laparoscopy; Instruments; minimally invasive surgery

STUDY DESIGN:
Intervention Model Description: prospective randomized trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be unaware that they will undergo an abdominal hysterectomy using VCare or SecuFix for their surgical procedure.
  Data entry will utilize a coded system within a pre-designed SPSS spreadsheet. A research assistant, who will be independent of the intervention administration, will enter data for each patient using a designated code (1 or 2) that corresponded to the group assignment. All data will send to an independent statistician for blinded analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SecuFix UM (Experimental): SecuFix UM arm: patients undergoing total laparoscopic hysterectomy
  Interventions: Device: SecuFix UM
- VCare UM (Active Comparator): VCare UM arm: patients undergoing total laparoscopic hysterectomy
  Interventions: Device: VCare UM

INTERVENTIONS:
Device: SecuFix UM — All surgeries were performed using Secufix UM.
  Arms: SecuFix UM
Device: VCare UM — All surgeries were performed using VCare UM.
  Arms: VCare UM

SUMMARY:
Hysterectomy, the most commonly performed gynecological operation, can be carried out through various methods using a wide array of instruments and energy techniques. Minimally invasive procedures such as robotic or laparoscopic approaches are linked to lower perioperative complications and quicker recovery when compared to abdominal hysterectomy. Furthermore, recent advancements in surgical tools and methodologies have facilitated endoscopic surgeries. Uterine manipulation plays a crucial role in laparoscopic hysterectomy by facilitating bladder dissection, positioning the ureters, and exposing the anterior and posterior vaginal fornices. It also prevents pneumoperitoneum loss by closing off the vaginal space. Despite these apparent benefits, there is no existing report comparing different types of uterine manipulators. Therefore, the purpose of this study was to compare the Vcare and SecuFix uterine manipulators used in laparoscopic hysterectomy based on operative time, length of hospital stay, estimated blood loss, perioperative complications, and subjective performance.

DETAILED DESCRIPTION:
Introduction Hysterectomy is the most commonly performed gynecological operation and can be carried out through various methods using a wide array of instruments and energy techniques. Although the methods have advantages and disadvantages over each other, minimally invasive procedures are associated with less morbidity and perioperative recovery. Recent advancements in surgical tools and methodologies have facilitated endoscopic surgeries. Uterine manipulation is crucial in laparoscopic hysterectomy as it facilitates bladder dissection, positioning the ureters, and exposing the anterior and posterior vaginal fornices. It also maintains pneumoperitoneum. Currently, many uterine manipulators are available, but the evidence for their efficacy and safety is still unclear. The purpose of utilizing a uterine manipulator is to enhance surgical outcomes and reduce intraoperative complications, particularly concerning the bladder and ureter. It is important to visualize the anterior and posterior fornices and ensure maintenance of the pneumoperitoneum. Therefore, uterine manipulators play a crucial role in laparoscopic hysterectomy. However, none of the manipulators currently available possess all the characteristics of an ideal manipulator. Therefore, the investigators aimed to compare the Vcare and SecuFix uterine manipulators used in laparoscopic hysterectomy with regard to operative time, length of hospital stay, estimated blood loss, and perioperative complications.

ELIGIBILITY:
Inclusion Criteria:

* aged 35-65 years
* hysterectomy for benign gynecological indications

Exclusion Criteria:

* history of urogynecologic procedures
* suspected gynecological malignancy,
* endometriosis,
* pelvic inflammatory disease,
* pelvic organ prolapse,
* unavailibility of operative records

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
operative time | Operation time was defined as the duration in minutes from the skin incision to detachment of the uterus during surgery.
  Operation time was defined as the duration from the skin incision to detachment of the uterus.

IPD SHARING:
Plan to Share IPD: No
The dataset used and/or analyzed in the study are available from the corresponding author on reasonable request.